CLINICAL TRIAL: NCT02724124
Title: Acute Effect of Static Stretching and Muscle Warming on the Functional Performance of College Volleyball Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Germanna de Medeiros Barbosa, physical therapist master; PhD student, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1.378.698
Record Dates: First submitted 2016-02-18; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Neuromuscular Manifestations
Keywords: exercise muscle stretching; electromyography
MeSH Terms: conditions — Neuromuscular Manifestations | interventions — Muscle Stretching Exercises; Warm-Up Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- static stretching (Experimental): group of 11 volunteers (gSS)
  Interventions: Other: Static Stretching
- warm up - (Experimental): group of 11 volunteers (gWU)
  Interventions: Other: warm up
- static stretching + warm up (Experimental): (group of 11 volunteers - SS+WU)
  Interventions: Other: static stretching + warm up
- warm up+static stretching (Experimental): (group of 11 volunteers - WU+SS)
  Interventions: Other: warm up+static stretching
- Control Group (Other): No intervention - athletes rested
  Interventions: Other: Control

INTERVENTIONS:
Other: Static Stretching — 3 sets of 30-second self static hamstring stretch (IT), quadriceps (QD) and sural triceps (TS) of both lower limbs, with an interval of 30 seconds of rest between sets
  Arms: static stretching
Other: warm up — Warm-up for 10 minutes at 70-80% of maximum heart rate.
  Arms: warm up -
Other: static stretching + warm up — 3 sets of 30-second self static hamstring stretch (IT), quadriceps (QD) and sural triceps (TS) of both lower limbs, with an interval of 30 seconds of rest between sets + Warm-up for 10 minutes at 70-80% of maximum heart rate.
  Arms: static stretching + warm up
Other: warm up+static stretching — Warm-up for 10 minutes at 70-80% of maximum heart rate + 3 sets of 30-second self static hamstring stretch (IT), quadriceps (QD) and sural triceps (TS) of both lower limbs, with an interval of 30 seconds of rest between sets
  Arms: warm up+static stretching
Other: Control — No intervention
  Arms: Control Group

SUMMARY:
The purpose of this study is analyze the effects of static stretching and active warm up, isolated and associated, in functional performance of the lower limbs in college volleyball athletes.

Study hypothesis:

H0: The stretching and / or warm up, alone or in combination, do not alter the functional performance of volleyball players.

H1: The stretching and / or warm up, alone or in combination, alter the functional performance of volleyball players.

DETAILED DESCRIPTION:
This is a cross-over study containing 11 volleyball athletes randomly divided into 5 groups: control (C), warming-up (gAQ), stretching (gAL), warming-up and stretching (gAQAL), stretching and warming-up (gALAQ). All subjects underwent the evaluation measures of functional performance that were conducted pre and post intervention.

ELIGIBILITY:
Inclusion Criteria:

1. being male;
2. were aged between 18 and 28 years of age;
3. no previous history of orthopedic disorders, rheumatic disorders, cardiovascular, metabolic and / or vestibular and neurological disorders that prevent them from participating in the study dysfunctions;
4. no history of injury, trauma or disease in the lower limbs in the last six months, without surgery;
5. participate in the University Selection UFRN;
6. training time display mode in the above two years with a frequency of at least three times a week.

Exclusion Criteria:

1. presence of injury during the survey period;
2. not conduct evaluative and intervention procedures;
3. waiver to participate.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Muscle Power | Evaluation of power after fifteen minutes the application of intervention
  Power measured by Jump System

IPD SHARING:
Plan to Share IPD: Yes
Each individual receives a report of their performance